CLINICAL TRIAL: NCT06601361
Title: Studying Non Alcoholic Fatty Liver Disease and Liver Fibrosis Among Systemic Lupus Erythematosus Patients At Assiut University Hospital
Acronym: NAFLD and SLE
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayman Makram Ayad Souliman, physician, Assiut University
Other Study IDs: NAFLD in SLE
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: NAFLD - Nonalcoholic Fatty Liver Disease
Keywords: NAFLD and SLE
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Fibroscan — Fibroscan (transient elastography ) is a non-invasive imaging method that evaluates steatosis and fibrosis by measuring liver stiffness using ultrasonographic sound waves. It is an acceptable alternative to liver biopsy and is fast , reliable, and reproducible, enabling screening and disease follow-up.11 It is now widely used to assess liver fibrosis in various liver diseases; however, currently there is no data on Fibroscan assessment regarding hepatic involvement in SLE patients. The aim of this study was to evaluate fatty liver and liver fibrosis in SLE patients using fibroscan and determine associated factors such as immunosuppressive medications.

SUMMARY:
Aim of the study :-

1. to estimate prevalence of non alcoholic fatty liver disease and liver fibrosis among Systemic lupus erythematosus patients
2. to determine risk factors in SLE patients contributing to NAFLD and liver fibrosis

DETAILED DESCRIPTION:
Lupus Erythematosus (SLE) is a systemic, multi organ, Autoimmune disease that more common in women than men and is typically diagnosed during the reproductive age .1 Lupus affects almost all organs and can present with awide variety of symptoms . Renal and skin involvement are the most frequently encountered presentation ,however gastrointestinal involvement is also seen in patients with SLE.2 involvement of liver in SLE is rare and mostly presents as asymptomatic hepatomegaly subclinical adiposity, and/or increased liver enzymes.3.4 Elevated transaminase levels may be observed in 15-55% of the patient population and can be associated with disease activity.4,5 The most common causes are drug-related liver injury (31%), lupus-associated hepatitis (29%), and fatty liver disease (18%).6 drugs used in the treatment of SLE patient such as non-steroidal anti-inflammatory drugs, glucocorticoids, cyclophosphamide ,mycophenolate mofetil, azathioprine, and methotrexate can all cause hepatotoxicity.7 As such, it is important to differentiate the etiology and determine whether hepatotoxicity is due to the medications used or the disease itself.

Non-alcoholic fatty liver disease (NAFLD) and liver fibrosis may both progress to cirrhosis and cause liver failure. NAFLD is also a risk factor for cardiovascular disease in the general population, which is also one of the most important causes of morbidity and mortality in lupus patients.8,9 Even though hepatomegaly and hepatosteatosis are frequently observed in abdominal imaging performed for other reasons in SLE patients, the majority of these cases are not evaluated further since the gold standard for diagnosis is liver biopsy, an invasive procedure associated with a number of serious complications.10 Therefore, the prognostic significance of NAFLD and liver fibrosis is still largerly unknown in these patients.

Fibroscan (transient elastography ) is a non-invasive imaging method that evaluates steatosis and fibrosis by measuring liver stiffness using ultrasonographic sound waves. It is an acceptable alternative to liver biopsy and is fast , reliable, and reproducible, enabling screening and disease follow-up.11 It is now widely used to assess liver fibrosis in various liver diseases; however, currently there is no data on Fibroscan assessment regarding hepatic involvement in SLE patients. The aim of this study was to evaluate fatty liver and liver fibrosis in SLE patients using fibroscan and determine associated factors such as immunosuppressive medications.

.Several non-invasive diagnostic scores for non-alcoholic fatty liver (NAFL) have been developed one of the most recent scores is HSI score hepatic steatosis index Multivariate analysis indicated that high serum alanine aminotransferase (ALT) to serum aspartate aminotransferase (AST) ratio, high body mass index (BMI), and diabetes mellitus were independent risk factors of NAFLD (all P < 0.001). Using these variables, a formula was derived by a logistic regression model: hepatic steatosis index (HSI) = 8 × (ALT/AST ratio) + BMI (+2, if female; +2, if diabetes mellitus). HSI had an area under receiver-operating curve of 0.812 (95% confidence interval, 0.801-0.824). At values of <30.0 or >36.0, HSI ruled out NAFLD with a sensitivity of 93.1%, or detected NAFLD with a specificity of 92.4%, respectively. Of 2692 subjects with HSI <30.0 or >36.0 in the derivation cohort, 2305 (85.6%) were correctly classified. HSI was validated in the subsequent validation cohort.

HSI is a simple, efficient screening tool for NAFLD that may be utilized for selecting individuals for liver ultrasonography and for determining the need for lifestyle modifications.12

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years old ,Both sex male and female, diagnosed with SLE

Exclusion Criteria:

1. Age below 18 years old
2. patients with hepatitis b virus (HBV), hepatitis c virus (HCV) or cirrhosis
3. malignancy, cardiac disease,
4. patients on dialysis.
5. obese patient, BMI more than 30

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 years old ,Both sex male and female, diagnosed with SLE
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
estimation of prevalence of non alcoholic fatty liver disease and liver fibrosis among Systemic lupus erythematosus patients | baseline
  We will divide lupus patients into 3 groups group number 1 who are SLE patient in activity and not taking treatment,group number 2 who are SLE patients in activity and taking treatment and controlled,group number 3 who are SLE patients in activity and taking treatment but not controlled our outcome is to estimate prevalence of NAFLD in each group .

SECONDARY OUTCOMES:
determinate risk factors in SLE patients contributing to NAFLD and liver fibrosis | baseline
  We will determine the risk factor in SLE patients we take and determine the risk factors in patients detected as having NAFLD and determine the risk factors may contributed to develop NAFLD

REFERENCES:
- [Background] Yetginoglu O, Atas DB, Yilmaz Y, Velioglu A, Arikan H, Alibaz-Oner F, Direskeneli H, Tuglular S, Asicioglu E. Fibroscan detection of fatty liver and liver fibrosis in patients with systemic lupus erythematosus. Lupus. 2022 May;31(6):723-729. doi: 10.1177/09612033221094708. Epub 2022 Apr 10. PMID 35403493